CLINICAL TRIAL: NCT06967623
Title: Comparison of the Effectiveness of Diaphragm Thickness in Indicating Weaning Success With Other Weaning Parameters in Patients Followed up in the Intensive Care ünit
Brief Title: Comparison of Weaning Parameters and Diaphragm Thickness Changes
Acronym: Weaning
Status: Completed | Type: Observational
Sponsor: Tarık Durna (Other)
Responsible Party: Sponsor-Investigator, Tarık Durna, Medical Doctor, Namik Kemal University
Organization: Namik Kemal University (Other)
Other Study IDs: 2022.111.06.01; tarık durna (Other: Namik Kemal University)
Record Dates: First submitted 2025-03-24; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Mechanical Ventilation; Weaning Failure; Intensive Care Unit (ICU) Patients; Diaphragm Dysfunction
Keywords: Diaphragm ultrasonography; Mechanical ventilation; Diaphragm thickness; Weaning; Weaning parameters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- weaning successful: Patients who can maintain spontaneous breathing for 48 hours
  Interventions: Device: diaphragm ultrasound
- weaning failed: Patients who have failed spontaneous breathing attempts or require intubation within 48 hours after extubation
  Interventions: Device: diaphragm ultrasound

INTERVENTIONS:
Device: diaphragm ultrasound — On the day of hospitalization or the first day of mechanical ventilation, the patient's position was elevated by 30°, and the high-frequency linear probe of the ultrasound was placed perpendicular to the skin in the cranio-caudal direction, and the diaphragm apposition zone, where the right anterior and middle axillary line corresponds to the 8th-10th intercostal space, was imaged and measurements were made with B mode.

SUMMARY:
Determining the appropriate timing for mechanical ventilator weaning in intensive care unit patients is critical to avoid complications related to early or late weaning, including weaning failure. Common predictors such as P0.1, F/VT, WOB, and P0.1 × F/VT are routinely used to guide this decision. Recently, diaphragm muscle weakness has been recognized as a significant contributor to weaning failure. Ultrasound has emerged as a useful, repeatable, and non-invasive tool for assessing diaphragmatic function.

This study investigates the relationship between ultrasound-based diaphragm thickness changes and standard weaning predictors. It also evaluates the impact of demographic variables such as age, gender, weight, and comorbidities on diaphragm thickness. A total of 68 mechanically ventilated patients, aged 18 years or older, with Glasgow Coma Scale >8 and BMI <35, were included. Ultrasound measurements were performed on the first day of intubation and prior to extubation, using a high-frequency linear probe from the right anterior mid-axillary line at the 8th-10th rib level. Weaning was considered successful if patients maintained spontaneous breathing for 48 hours post-extubation.

DETAILED DESCRIPTION:
Study Title: The Relationship between Diaphragm Thickness Changes and Weaning Predictors in Intensive Care Unit Patients on Mechanical Ventilation

Background: Mechanical ventilation weaning, or transitioning patients from mechanical ventilators to spontaneous breathing, is a critical step in intensive care. The decision on the optimal timing of weaning is pivotal for patient recovery and minimizing complications. Early or delayed weaning may lead to failure, which significantly increases mortality and morbidity rates. Traditional weaning predictors such as P0.1, F/VT, WOB, and P0.1 X F/VT are widely used in intensive care units (ICUs), but none provide a comprehensive assessment of diaphragmatic function.

Recent studies have indicated diaphragm weakness as a potential major cause of weaning failure, and ultrasonography of the diaphragm has gained attention as a practical, reliable, and cost-effective diagnostic tool. Given its growing popularity, we aimed to assess the relationship between changes in diaphragm thickness-measured using ultrasound-and conventional weaning predictors in ICU patients.

Study Objective: The primary goal of the study was to observe the relationship between diaphragm thickness changes and conventional weaning parameters. Additionally, the study aimed to statistically investigate the effects of demographic variables such as age, gender, weight, and comorbidities on diaphragm thickness change and its potential implications for weaning success.

Methodology:

Study Design: A prospective observational study.

Study Population: 68 ICU patients, aged 18 years or older, who were intubated, had a Glasgow Coma Scale higher than 8, and had been on mechanical ventilation for at least 24 hours. Patients with a BMI greater than 35 were excluded.

Inclusion Criteria: Patients who met the weaning criteria and who had consented to participate in the study.

Exclusion Criteria: Patients with major contraindications to ultrasound (e.g., open chest surgery), or those with known neuromuscular disorders.

Ultrasonographic Measurements: On the first day of intubation or admission, diaphragm thickness was measured at the 8th and 10th ribs from the right anterior mid-axillary line using a high-frequency linear probe in B mode. Three repetitions were performed for each measurement, and the average was recorded. The second diaphragm thickness measurement was taken just before extubation in patients assessed as suitable for weaning.

Weaning Process: Weaning was attempted in patients who met routine criteria, including stable respiratory parameters (RSBI, P0.1, WOB, etc.). After weaning, the patients were extubated and observed for 48 hours. Those who maintained spontaneous breathing were considered successful weaning cases, while those who required reintubation were categorized as weaning failures.

Statistical Analysis: The statistical analysis focused on comparing the initial and final diaphragm thickness between the weaning success and failure groups. Additionally, the correlation between diaphragm thickness change and the duration of mechanical ventilation was explored. Multivariate regression models were used to adjust for potential confounding factors, including age, gender, weight, and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants aged 18 years or older.
* Intubation Status: Participants who are intubated and receiving mechanical ventilation for at least 24 hours.
* Glasgow Coma Scale (GCS): Participants with a GCS score of greater than 8 at the time of enrollment.
* Body Mass Index (BMI): Participants with a BMI lower than 35.
* Weaning Suitability: Participants who are being evaluated for weaning from mechanical ventilation based on routine ICU weaning parameters.
* Informed Consent: Participants or their legal representatives must provide informed consent to participate in the study.

Exclusion Criteria:

* Age: Participants younger than 18 years.
* Neurological or Cognitive Impairments: Participants with neurological or cognitive conditions that may affect the ability to participate in the study or give informed consent.
* Mechanical Ventilation Duration: Participants who have been on mechanical ventilation for less than 24 hours at the time of enrollment.
* Severe Respiratory Conditions: Participants with conditions such as acute respiratory distress syndrome (ARDS) or those requiring higher levels of respiratory support, such as invasive or non-invasive positive pressure ventilation.
* Severe Heart Failure: Participants with severe heart failure or other critical cardiovascular conditions that may interfere with the ability to tolerate weaning procedures.
* Pregnancy: Female participants who are pregnant or breastfeeding.
* Other Contraindications: Any participant for whom diaphragm ultrasound measurements would be technically difficult or clinically inappropriate (e.g., due to anatomical or technical factors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 68 adult participants (18+ years) who are intubated and undergoing mechanical ventilation for at least 24 hours in an ICU. Inclusion Criteria: Intubated for 24+ hours, Glasgow Coma Scale (GCS) > 8, BMI < 35, meets weaning criteria, willing to consent. Exclusion Criteria: Age < 18, severe cognitive or neurological impairment, ventilation < 24 hours, severe comorbidities, pregnancy/breastfeeding, contraindications for diaphragm ultrasound. Population Characteristics: The cohort will consist of ICU patients being evaluated for weaning, representing a range of ages, genders, and comorbidities. Demographic and clinical data will be analyzed for correlations with diaphragm thickness change and weaning success. Study Design: An observational cohort study using ultrasound to assess diaphragm thickness in relation to mechanical ventilation weaning outcomes.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Diaphragm Thickness | From Day 1 of mechanical ventilation to the day of planned extubation, up to 14 days
  The primary outcome of the study will be the change in diaphragm thickness, measured using ultrasound before and after extubation.
Number of Participants with Successful Weaning (Maintaining Spontaneous Breathing for ≥48 Hours Post-Extubation) | Up to 48 hours after extubation
  Weaning success will be defined as the patient's ability to maintain spontaneous breathing without the need for reintubation or mechanical ventilatory support for at least 48 hours following extubation. Participants who require reintubation or ventilatory assistance within 48 hours will be considered as weaning failures.

CONTACTS AND LOCATIONS:
Locations (1):
- Namık Kemal University Hospital, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) with other researchers. Access to the data will be restricted to the study team for the purposes of this research only, in compliance with ethical and regulatory guidelines.